CLINICAL TRIAL: NCT04996719
Title: Effect of Rapamycin to Improve Cardiac Function in Frail Older Adults With Heart Failure With Preserved Ejection Fraction: A Randomized Pilot and Proof-of-Concept Study
Brief Title: Effect of Rapamycin to Improve Cardiac Function in Frail Older Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Mandeep Singh, Professor of Medicine, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-003837
Record Dates: First submitted 2021-08-03; First posted 2021-08-09 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Rapamycin (Experimental): find safe doses for patients who have heart failure with preserved ejection fraction
  Interventions: Drug: Rapamune

INTERVENTIONS:
Drug: Rapamune — We will start the dose at 0.5mg capsule every other day for 2 weeks. If participants tolerate this dose and trough blood levels are (≤4ng/mL), the dose of rapamycin will be increased to 0.5mg daily for the duration of the study. If necessary, dose can remain at 0.5 mg every other day, depending on the trough level. To avoid immunosuppression, we will target lower dose of rapamycin, maintain lower trough serum levels (≤4ng/mL).
  Other Names: Rapamycin

SUMMARY:
The purpose of this research is to see if the drug rapamycin will improve the heart's ability to pump by improving your oxygen consumption.

DETAILED DESCRIPTION:
This will be a pilot, proof-of-concept study. Patients 60 years or older with invasively proven HFpEF or have definite HFpEF as determined by the 2 established scores and frailty (positive screen for computable phenotype), will be approached for enrollment. Subjects meeting screening criteria following written informed consent will be randomized to receive rapamycin or matching placebo (study drug). Efficacy outcomes will be measured at baseline and at 6 months. Safety will be assessed by in person or remote video monitoring weekly for 1 month, then monthly for 5 months till the end of the study. We will also measure trough rapamycin levels (≤4ng/mL) twice-a-month for the first month and then monthly for 5 months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥60 years
* Diagnosis of HFpEF by either H2FEPF score of 6-9 or HFA-PEFF score of 5-6, or invasively confirmed diagnosis of HFpEF (resting pulmonary capillary wedge pressure ≥15mmHg or ≥25mmHg with exercise).
* Diagnosis of computable phenotype of frailty rests on screening questions about ability to climb two flights of stairs, activities of daily living, living environment, wearing of dentures/hearing aids, and whether the patient uses assistive devices.

Exclusion Criteria:

* Reduced ejection fraction (≤50%) with or without prior history of myocardial infarction
* Acute coronary syndrome <3 months
* Uncontrolled diabetes mellitus (HbA1C>8)
* Uncontrolled hypertension (>160/100mmHg, despite 3 antihypertensive medications)
* Nephrotic syndrome or eGFR <30mL/min/1.73m2
* Cirrhosis
* Hepatitis B/C positive
* Elevated lived enzymes (AST/ALT>3ULN
* Prior malignancy other than basal cell carcinoma
* History of ongoing, chronic or recurrent infectious disease
* Suspected/proven immunocompromised state
* Uncontrolled hyperlipidemia (fasting TG >400 mg/dL (>4.5 mmol/L) or total cholesterol >300 mg/dL (>7.8 mmol/L) despite maximum lipid lowering therapy
* Class IV HF symptoms

Ages: 60 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-05-24 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2023-08-25 (Actual)

PRIMARY OUTCOMES:
Change cardiopulmonary reserve capacity by improving peak VO2 with rapamycin | 6 months
  In this pilot, proof-of-concept study, we hypothesize that in older adults (≥60 years) with HFpEF who are frail, chronic rapamycin administration will change their cardiopulmonary reserve capacity by improving peak VO2.Primary safety objective is the safety of rapamycin.

CONTACTS AND LOCATIONS:
Overall Officials: Mandeep Singh, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials